CLINICAL TRIAL: NCT06963359
Title: Preventing Loss of Autonomy in Older Patients by Improving Diagnosis of Sarcopenia and Monitoring With High-definition Surface Electromyography Technology
Brief Title: High-definition Surface Electromyography Markers for the Diagnosis and Monitoring of Sarcopenia
Acronym: CHRONOSSARCRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Compiègne University of Technology (Unknown); Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP240022
Record Dates: First submitted 2024-01-12; First posted 2025-05-09 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Sarcopenia
Keywords: High definition surface electromyography; Sarcopenia; Muscle
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elderly patients suspected of sarcopenia (Experimental)
  Interventions: Device: HD-sEMG; Device: Quadriceps muscle ultrasound; Other: IPAQ Physical Activity Questionnaire

INTERVENTIONS:
Device: HD-sEMG — High definition surface electromyography, allowing the recording of muscle activation signals sensitive to the intensity of the contraction and indirectly to the muscle strength as well as to the muscular fatigability, but also capable of measuring the modifications of the recruitment modalities of the motor units. This recording will be made on the rectus femoris during knee extension, either in the lying position or during chair rises, depending on the patient's functional state
Device: Quadriceps muscle ultrasound — Muscle Ultrasound with Philips Lumify Wireless Handheld Ultrasound for Android - Model - L12-4 linear probe, allowing performance at the patient's bed
Other: IPAQ Physical Activity Questionnaire — Physical activity assessment questionnaire/adapted version for seniors

SUMMARY:
Sarcopenia is a progressive and generalised skeletal muscle disorder involving the accelerated loss of muscle mass and function that is associated with increased adverse outcomes including falls, functional decline, frailty, and mortality. In this project, the high-definition surface electromyography technology (HD-sEMG) signals will be analysed to extract features/ markers for the diagnosis of sarcopenia. This is a multicentric, descriptive, cross-sectional, parallel group study to develop a new diagnostic method.

It is planned to include 846 people aged 75 years and over hospitalized in the acute geriatric or rehabilitation wards and suspected of sarcopenia (Score ≥4 on the SARC-F screening questionnaire). The inclusion duration will be 18 months and adding a 3-month patient follow-up. The total study duration will be 21 months. Patients will have their body composition using bioimpedancemetry and if possible by dual X-ray absorptiometry (DEXA). Muscular strength will be assessed by handgrip strength. Physical performance will be assessed. Additional data will be collected from their medical records.

DETAILED DESCRIPTION:
The aging of the population is a major public health problem with its multifactorial impact on quality of life and maintenance of autonomy. Unfortunately, one consequence of aging is sarcopenia, which affects the intrinsic and functional properties of muscle. It is a risk factor for loss of autonomy, falls, frailty and is associated with increased mortality. Sarcopenia is defined as a progressive loss of muscle mass, strength and physical performance. Classically, sarcopenia is assessed by imaging techniques (MRI, DEXA) or bioelectrical impedancemetry for aspects related to the assessment of muscle mass loss. MRI or DEXA are not widely available and/or access is limited. For functional aspects, grip strength measurements are often used. Currently sarcopenia cannot be diagnosed and evaluated by a single examination, including both the morphological (muscle mass) and functional aspects. Furthermore, several biological markers are associated with muscle mass, strength, and function, but these biomarkers are not specific to skeletal muscle and are weakly associated with clinical goals. Finally, despite the important interest in assessing the qualitative/functional and quantitative aspect of skeletal muscle in neuromuscular impairment, there is currently no tool that routinely assesses these aspects. In this context, developing new approaches for non-invasive assessment of sarcopenia, is a major issue. In this project, the investigators aim to develop an automatic procedure derived from high-definition surface electromyography (HD-sEMG) technology, non-invasive and portable, for the diagnosis of sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 75 years and over
* Score ≥4 on the SARC-F screening questionnaire
* Enrolled in a social security plan (no AME)
* Informed and consenting patient

Exclusion Criteria:

* BMI ≥30 kg/m2
* Severe psychiatric pathology or severe cognitive disorders that do not allow the performance of examinations
* Patients who are dependent for all acts of daily life
* Patients with a very short life expectancy <3months
* Pace maker
* Recent fracture or trauma of the preventing dynamic measurement of HD-sEMG recording
* Bilateral hip prosthesis
* Skin problem that may interfere with the recording of surface EMG activity
* Skin allergies to plasters
* Allergies to electrode materials (acrylate)
* Patient under legal protection
* Patient on state medical aid (AME : Aide Médicale d'Etat)

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 846 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Diagnostic score of electromyographic signals from the rectus femoris collected by the HD-sEMG technique, differentiating sarcopenic from non-sarcopenic elderly subjects | Day 1- Day 7

SECONDARY OUTCOMES:
HD-sEMG signals associated with functional recovery | Day 21 +/-3 days
  Identify HD-sEMG parameters associated with good functional recovery of autonomy at D21 and M3 of hospitalization (muscle resilience)
HD-sEMG signals associated with functional recovery | Day 90+/-7 days
  Identify HD-sEMG parameters associated with good functional recovery of autonomy at D21 and M3 of hospitalization (muscle resilience)
HD-sEMG signals associated with Muscle Mass Index | Day 1
  Correlation between electromyographic signals from the rectus femoris collected using the HD-sEMG technique and the Muscle Mass Index measured by DEXA or Bioimpedancemetry
HD-sEMG signals associated with Muscle Mass Index | Day 7
  Correlation between electromyographic signals from the rectus femoris collected using the HD-sEMG technique and the Muscle Mass Index measured by DEXA or Bioimpedancemetry
HD-sEMG signals associated with grip strength | Day 1
  Correlation between electromyographic signals from the rectus femoris collected using the HD-sEMG technique and grip strength measured using manual hydraulic dynamometer
HD-sEMG signals associated with grip strength | Day 7
  Correlation between electromyographic signals from the rectus femoris collected using the HD-sEMG technique and grip strength measured using manual hydraulic dynamometer
HD-sEMG signals associated with physical performance | Day 1
  Correlation between electromyographic signals from the rectus femoris collected using the HD-sEMG technique and the physical performance measured using Short Physical Performance Battery score (bad physical performance if score ≤ 8).
HD-sEMG signals associated with physical performance | Day 7
  Correlation between electromyographic signals from the rectus femoris collected using the HD-sEMG technique and the physical performance measured using Short Physical Performance Battery score (bad physical performance if score ≤ 8).
HD-sEMG signals associated with quadriceps muscle and subcutaneous fat thickness | Day 1
  Correlation between electromyographic signals from the rectus femoris collected using the HD-sEMG technique and quadriceps muscle and subcutaneous fat thickness measured using portable ultrasound).
HD-sEMG signals associated with quadriceps muscle and subcutaneous fat thickness | Day 7
  Correlation between electromyographic signals from the rectus femoris collected using the HD-sEMG technique and quadriceps muscle and subcutaneous fat thickness measured using portable ultrasound).
Progress in muscle parameters | Day 21 +/-3 days
  Changes in muscle parameters mentioned above, between the D0 and D21.
Correlation between muscle parameters and in-hospital complications | Day 21 +/-3 days
  Study the relationship between muscle parameters and in-hospital complications. (cardiovascular, pulmonary and thromboembolic diseases)
Correlation between muscle parameters and quality of life | Day 1
  Study the relationship between muscle parameters and quality of life measured using EQD5 scale (EuroQol-5D; 0-20: higher scores mean a worse outcome).
Correlation between muscle parameters and quality of life | Day 21 +/-3 days
  Study the relationship between muscle parameters and quality of life measured using EQD5 scale (EuroQol-5D; 0-20: higher scores mean a worse outcome).
Correlation between muscle parameters and quality of life | Day 90+/-7 days
  Study the relationship between muscle parameters and quality of life measured using EQD5 scale (EuroQol-5D; 0-20: higher scores mean a worse outcome).

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Hôpital Corentin Celton, APHP, Issy-les-Moulineaux
  - Hôpital Charles Foix, APHP, Ivry-sur-Seine
  - Unité d'Explorations fonctionnelles du sujet âgé - Hôpital Charles Foix, Ivry-sur-Seine
  - Hôpital Rothschild, APHP, Paris
  - Hôpital Tenon, APHP, Paris

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.